CLINICAL TRIAL: NCT02317458
Title: EFFICACY AND SAFETY OF BONE MARROW-DERIVED MESENCHYMAL CARDIOPOIETIC CELLS (C3BS-CQR-1) FOR THE TREATMENT OF CHRONIC ISCHEMIC HEART FAILURE
Brief Title: Congestive Heart Failure Cardiopoietic Regenerative Therapy (CHART-2) Trial - THE CHART-2 TRIAL
Acronym: CHART-2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Celyad Oncology SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C3BS-C-12-01
Record Dates: First submitted 2014-12-09; First posted 2014-12-16 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active arm (Experimental): One arm with standard of care and C3BS-CQR-1 injection (treatment group) using intramyocardial catheter injection.
  Interventions: Biological: Experimental
- Control arm (Sham Comparator): One arm with standard of care undergoing a sham procedure (control group)using intramyocardial catheter injection. .
  Interventions: Biological: Sham comparator

INTERVENTIONS:
Biological: Experimental — One active arm with standard of car and treatment with C3BR-CQR-1 using intramyocardial injection
  Other Names: C3BR-CQR-1
  Arms: Active arm
Biological: Sham comparator — One arm with standard of care undergoing a sham procedure
  Arms: Control arm

SUMMARY:
This study is designed to evaluate the efficacy and safety of the C3BS-CQR-1 in the treatment of patients with chronic heart failure secondary to ischemic cardiomyopathy.

DETAILED DESCRIPTION:
Patients with chronic heart failure secondary to ischemic cardiomyopathy being on standard of care will be screened per the protocol inclusion and exclusion criteria. Enrolled patients will be randomized on a 1:1 ratio to either standard of care and C3BS-CQR-1 injection (treatment group) or standard of care undergoing a sham procedure (control group). Patients randomized to the treatment group, for which C3BS-CQR-1 production met release criteria, will undergo endoventricular injection of the C3BS-CQR-1 using injection catheter.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and < 80 years.
2. Systolic dysfunction with LVEF ≤ 35% as assessed by echocardiography.
3. Ischemic heart failure ineligible for further revascularization. Ischemic heart failure is defined as history of myocardial infarction or evidence of clinically significant coronary disease associated with LV systolic dysfunction leading to HF. The patient must not be a candidate for revascularization in the judgment of the investigator, based on the absence of unstable coronary-related symptoms and either non-invasive testing or coronary angiography within 24 months prior to screening.
4. Total MLHFQ score > 30.
5. Ability to perform a Six-Minute Walk Test > 100 m and ≤ 375 m.
6. History of hospitalization for HF within 12 months prior to screening or treatment in an out-patient clinic with intravenous therapy (including vasodilators, positive inotropic agents, vasopressors or diuretics) for worsening HF within 12 months prior to screening. Be or must have been diagnosed within the previous 12 months in NYHA class III or IV or INTERMACS class 4, 5, 6 or 7, and at the time of inclusion, must be at least in NYHA class II or greater. If in NYHA class II, 2 or more HF worsening events or NT-ProBNP > 1000 pg/mL requiring hospitalization or outpatient IV therapy during the prior 12 months are required.
7. Use of ACE inhibitor and/or ARB or sacubitril/valsartan (Entresto™); and beta blocker, for at least 3 months prior to screening visit, unless intolerant or contraindicated.
8. Stable dosing of ACE inhibitor or ARB or sacubitril/valsartan (Entresto™) and beta blocker, aldosterone blocker, and diuretics for at least one month prior to screening visit, defined as ≤50% change in total dose of each agent.
9. Willing and able to give written informed consent.

Exclusion Criteria:

1. Women who are pregnant, confirmed by a positive urine or serum hCG laboratory test at screening.
2. Women of child-bearing potential without a negative serum or urine pregnancy test at screening or who are not practicing a reliable form of birth control. Women who are postmenopausal (12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH level > 40 mIU/mL or 6 weeks post-surgical bilateral oophorectomy) or surgically sterile are not considered to be of child-bearing potential. Reliable contraception includes surgical sterilization, hormonal contraception, or double-barrier methods.
3. Men refusing to exercise a reliable form of contraception unless partner is unable to conceive.
4. Acute coronary syndrome leading to myocardial infarction or unstable angina within 90 days of screening.
5. Percutaneous coronary intervention (PCI) within 90 days prior to screening, or CABG surgery within 180 days prior to screening.
6. Patient on a cardiac transplant list or previously received any solid organ transplant.
7. Previously underwent cardiac surgery with remodeling procedure, left ventricular assist device placement or cardiomyoplasty. This exclusion does not apply to patients who underwent ventricularplasty without placements device >1 year ago.
8. Patient has undergone cardiac resynchronization therapy (CRT) within 6 months (180 days) prior to screening.
9. Severe uncontrolled HF requiring need for intravenous diuretics or inotropic support within 1 month prior to screening.
10. Inability to perform a Six-Minute Walk Test due to physical limitations other than HF including:

    1. Severe peripheral vascular disease
    2. Severe pulmonary disease or chronic obstructive pulmonary disease (COPD) with FEV1 <30% predicted
    3. Orthopedic limitations, severe muscular diseases, any other joint or muscular disease or neurological disorder (such as an old stroke or neuropathy) limiting the ability to walk for 6 minutes.
11. Dependence on chronic oral steroid therapy.
12. Stroke or transient ischemic attack leading to limitations in lower extremities or occurring within 180 days prior to screening.
13. Active myocarditis, constrictive pericarditis, restrictive, hypertrophic or congenital cardiomyopathy.
14. BMI < 19 or > 40 kg/m2.
15. Left ventricular thrombus.
16. Left ventricular wall thickness < 8mm visualized in more than 50% of LV, and defined as a "LV no-go zone
17. LV aneurysm or candidate for surgical aneurysmectomy.
18. Sustained VT or VF which led to AICD therapy (shock) within 3 months prior to screening.
19. Primary valvular disease of ≥ moderate degree, including mitral or aortic stenosis (with aortic valve area < 1.5 cm2) or regurgitation. Secondary mitral and tricuspid regurgitation due to LV dilatation will not be excluded
20. Prosthetic valve in aortic or mitral position, or prior MitraClip placement.
21. Chronic infection or active malignancy.
22. Compromised renal function as reflected by a serum creatinine level >2,0 mg/dL (>0.177 mmol/l) or is currently on dialysis.
23. Hematocrit < 28%.
24. Atherosclerosis and/or tortuosity of the aorta, iliac or femoral arteries of a degree that could impede or preclude the safe retrograde passage of the delivery catheter, including untreated aneurysm of the aorta.
25. Chronic immunosuppressive therapy due to inflammatory or systemic disease.
26. Patient tested positive for HIV 1 or 2, Hepatitis B or C, HTLV 1 or syphilis (as detailed in Section 19.1).
27. Exposure to any previous experimental cell or angiogenic therapy and/or myocardial laser therapy and/or therapy with another investigational drug within 60 days prior to screening or enrollment in any concurrent study that may confound the results of this study.
28. Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or in the opinion of the investigator are not suitable to participate.
29. Any illness other than CHF which might reduce life expectancy to less than 2 years from screening.
30. Known and relevant allergies and/or hyper-sensitivities to Dextran or other plasma volume expanders (including Gentran, Hyskon and Macrodex), to Bovine Serum Albumin (BSA) or to any albumin from animal origin.
31. Known severe allergy to the cardiac radiological contrast mixture.
32. Required dosage of cardiopoietic cells not reached

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-06; Primary Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of C3BS-CQR-1 injection based on a hierarchical composite score | 52 weeks
  1. Died of CV cause
  2. Hospitalized 2 or more times for HF
  3. Hospitalized once for HF
  4. Minnesota Living with Heart Failure Questionnaire (MLHFQ) total score worsened by 10 or more points
  5. MLHFQ total score neither worsened by 10 or more points nor improved by 10 or more points, or died of non-CV cause
  6. MLHFQ total score improved by 10 or more points